CLINICAL TRIAL: NCT01637649
Title: Diaphragm Function Evaluation in Stroke Patients During Voluntary Cough Using Sonography
Brief Title: Diaphragmatic Function in Stroke Patients.
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Sun Im, Assistant Professor, The Catholic University of Korea
Other Study IDs: 5-2-0120-60-668
Record Dates: First submitted 2012-07-07; First posted 2012-07-11 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Paralytic Stroke; Cough
Keywords: dysphagia,diaphragm, ultrasonography, inspiration, expiration,
MeSH Terms: conditions — Stroke; Cough; Deglutition Disorders; Respiratory Aspiration; Death

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Stroke patients with dysphagia: Stroke patients with confirmed evidence of aspiration and severe dysphagia tha would require modified diet or nasogastric tube feeding
- Stroke patients without dysphagia: Stroke patients but with no gross evidence of dysphagia or with mild dysphagia with a Penetration aspiration scale of less than 4
- healthy volunteer group: healthy volunteers with no prior history of dysphagia or stroke and who are not included in the exclusion criteria

SUMMARY:
* This study attempts to elucidate whether stroke patients with dysphagia have reduced diaphragm movement during voluntary coughing, and also during deep inspiration and expiration than stroke patients without dysphagia.
* This study will also compare various spirometric measurements with the diaphragmatic motions.

DETAILED DESCRIPTION:
Stroke is a debilitating condition that can impair multiple functions, including swallowing. Stroke patients with dysphagia, are known to have reduced cough due to multiple mechanisms and this can impair their expectorate function. This can lead to accumulation of sputum and mucoid, ultimately resulting in aspiration pneumonia. Stroke patients, especially those with dysphagia, are also known to have expiratory muscle weakness and weak cough than healthy controls. Stroke patients are also known to have reduced diaphragm movement than healthy subjects. Sonography is a useful tool that can easily and reliability measure diaphragm movement. Whether stroke patients with dysphagia have reduced diaphragm movement than those without dysphagia and whether this affects voluntary cough have not been reported yet.

This study attempts to evaluate diaphragm movements during voluntary cough in stroke patients with dysphagia and determine whether this reduced diaphragm movement correlates to their peak flow meters during voluntary cough.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients with confirmed unilateral brain lesion
* Gross aspiration confirmed via FEES or VFSS that would require non oral feeding for group 1.
* No gross evidence of dysphagia that would require non oral feeding for group 2.
* No prior episode of stroke or dysphagia for the healthy control group.

Exclusion Criteria:

* Episode of acute pneumonia or pulmonary embolism at time of enrollment
* Previous history of chronic respiratory disorders or other systemic disorders that may affect respiratory function ( ex, rheumatoid arthritis, chronic renal disease, spinal cord injury)
* Stroke patients with multiple brain lesions
* Episode of Diaphragm weakness due to peripheral polyneuropathy or unilateral phrenic nerve palsy
* Previous episode of abdominal or thoracic surgery within one year of enrollment
* Concomitant diagnosis of myopathy, muscular dystrophy or other disorders that may affect respiratory muscles.
* Episode of rib fracture within one year of enrollment
* Chronic alcoholism
* Patient with previous diagnosis of dementia or with impaired cognitive function that may limit full participation at the evaluation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke patients from a university affiliated medical center
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Diaphragm movement during coughing | 1 day
  Diaphragm movement during voluntary coughing will be recorded by musculoskeletal sonogrpahy

SECONDARY OUTCOMES:
Maximal inspiratory and expiratory pressure | 1 day
  respiratory pressure meter would be used to measure inspiratory and expiratory strength
Pulmonary Function test | 1 day
  FVC, FEV1, FEF 25-75%, FVC/FEV1 ( % ), Peak cough flow
Motricity index | Baseline
Canadian Neurological Stroke Scale | Baseline
Diaphragm movement during inspiration | 1 day
  Diaphragm movement will be recorded after deep inspiration
Diaphragm movement during expiration | 1 day
  Diaphragm movement during expiration will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Sun Im, MD, PhD, Principal Investigator — Department of Rehabilitation Medicine, Bucheon St Mary's Hospital, Catholic University of Korea, College of medicine
Locations (1):
- Bucheon St Mary's Hospital, Catholic University of Korea, Bucheon-si, Gyenoggido, South Korea

REFERENCES:
- [Derived] Park GY, Kim SR, Kim YW, Jo KW, Lee EJ, Kim YM, Im S. Decreased diaphragm excursion in stroke patients with dysphagia as assessed by M-mode sonography. Arch Phys Med Rehabil. 2015 Jan;96(1):114-21. doi: 10.1016/j.apmr.2014.08.019. Epub 2014 Sep 16. PMID 25234476